CLINICAL TRIAL: NCT03766841
Title: Avoiding Health Disparities When Collecting Patient Contextual Data for Clinical Care and Pragmatic Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Bradley Crotty, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PRO00031177
Record Dates: First submitted 2018-11-29; First posted 2018-12-06 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Communication
Keywords: consumer informatics; communication; patient engagement
MeSH Terms: conditions — Communication; Patient Participation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitated Enrollment (Experimental): Patients will be aided in the account creation and usage of a consumer informatics tool to collect and report patient-contextual data within the electronic health record
  Interventions: Behavioral: Facilitated Enrollment
- Usual Care (No Intervention): Patients will be invited to use the patient contextual data tool as per usual care, but will not receive additional assistance in account creation and usage.

INTERVENTIONS:
Behavioral: Facilitated Enrollment — Research coordinator will assist patients in account creation and usage of the tool.
  Arms: Facilitated Enrollment

SUMMARY:
To assess whether the routine collection of patient-contextual data improves patient activation and communication, and can mitigate racial disparities in communication and engagement, we are inviting patients who have upcoming appointments at the participating health system to participate in a communication study. Patients will be randomized to having guided (facilitated) enrollment in a tool that collects patient contextual data, or to usual care. All patients are invited directly by the health system to use the tool. Statistical methods will be used to determine the impact of the tool's use on outcomes of interest, as well as the impact on completion by the use of the facilitated enrollment. The study will particularly focus on assessing the impact of patient-contextual data and communication on heath disparities.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older
* able to speak and understand English,
* a patient at a selected Froedtert & Medical College of Wisconson primary care or internal medicine clinic (i.e., General Internal Medicine On Campus of Milwaukee Regional Medical Center, Sargeant Health Center, or Tosa Health Center (Plank Road Clinic) with an upcoming (> 4 weeks away) appointment and at least 1 previous appointment with the same provider in the previous 12 months.
* Patients with cognitive impairment (e.g. dementia) are eligible to participate through the use of proxies who would ordinarily accompany them to appointments and complete forms or post-visit surveys on their behalf.

Exclusion Criteria:

* Minors and non-English speaking patients are not eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Composite Communication Score As Assessed by Communication Assessment Tool, a validated 14-item patient-reported outcome. | Post Visit ( 1 week)
  Use of Communication Assessment Tool (CAT), a 14-item instrument that reports patient-views of clinician communication Makoul G, Krupat E, Chang CH. Measuring patient views of physician communication skills: development and testing of the Communication Assessment Tool. Patient Educ Couns. 2007;67: 333-342.

SECONDARY OUTCOMES:
Change in the composite score of the patient activation measure, a validated instrument to assess a patient's engagement and activation in their health issues. | Pre/Post Visit (1 week)
  Short form developed by J Hibbard et al on patient activation Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005;40: 1918-1930.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley H Crotty, MD MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Holt JM, Cusatis R, Winn A, Asan O, Spanbauer C, Williams JS, Flynn KE, Somai M, Talsma A, Laud P, Makoul G, Crotty BH. Impact of Pre-visit Contextual Data Collection on Patient-Physician Communication and Patient Activation: a Randomized Trial. J Gen Intern Med. 2021 Nov;36(11):3321-3329. doi: 10.1007/s11606-020-06583-7. Epub 2021 Feb 9. PMID 33559067
- [Derived] Holt JM, Winn A, Cusatis R, Talsma A, Crotty BH. Racial Disparities in Patient Activation: The Role of Economic Diversity. West J Nurs Res. 2021 Jun;43(6):517-529. doi: 10.1177/0193945920963130. Epub 2020 Oct 5. PMID 33012264
- [Derived] Holt JM, Cusatis R, Winn A, Asan O, Spanbauer C, Williams JS, Flynn KE, Somai M, Laud P, Crotty BH. The Impact of Previsit Contextual Data Collection on Patient-Provider Communication and Patient Activation: Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Sep 23;9(9):e20309. doi: 10.2196/20309. PMID 32965223